CLINICAL TRIAL: NCT00375648
Title: Assessment of the Efficacy and Safety of Zoledronic Acid in the Treatment of Bone Metastases-related Pain in Patients With Prostate Cancer
Brief Title: Efficacy and Safety of Zoledronic Acid in the Treatment of Bone Metastases-related Pain in Patients With Prostate Cancer
Acronym: TRAPEZE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EFR08
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: Prostate; Cancer; Bone metastases; Zoledronic acid; Bone metastases-related pain; Prostate cancer
MeSH Terms: conditions — Pain; Neoplasms; Prostatic Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- zoledronate (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
This study will evaluate the efficacy and safety of 4 mg zoledronic acid administered intravenously every 3-4 weeks in the treatment of bone metastases-related pain in patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate
* Bone-scan documented metastases
* Age > 18 years
* Non-controlled bone pain despite systemic anti-tumor therapy (hormone or chemotherapy) initiated at least 4 weeks before inclusion
* Life expectancy > 3 months
* Written informed consent

Exclusion Criteria:

* New systemic anti-tumor therapy initiated less than 4 weeks before study entry or predictable need for starting a new treatment within 8 weeks
* Radiation therapy on bone target lesions or bone-targeted isotope therapy (strontium or samarium) completed less than 4 weeks before study entry
* Bisphosphonate therapy within 8 weeks before study entry
* Abnormal renal function (serum creatinine > 2 x the upper normal limit or creatinine clearance < 30 ml/min)
* Corrected serum calcium > 3 mmol/L or < 2 mmol/L
* Clinically relevant hypersensitivity to zoledronic acid, or another bisphosphonate, or one component present in the formulation of the study drug
* Severe concomitant medical condition that could hamper patient's quality of life or influence the interpretation of pain
* Patients unable to fill in a questionnaire (neurologic or psychiatric conditions, illiteracy, etc.)

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-06; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
to measure the intensity of the pain relief of the patients at the end of treatment with a five classes score (TOTPAR = TOTal PAin Relief) | at 12 weeks or at 16 weeks (end of treatment)

SECONDARY OUTCOMES:
To measure the intensity of the pain relief of the patients with the PAR at each visit | every 3 or 4 weeks during 12 to 16 weeks
To evaluate the pain variation with VAS between V1 and V2, V3, V4, V5. | every 3 or 4 weeks during 12 to 16 weeks
To evaluate the pain variation with BPI (=Brief Pain Inventory) and correlate with VAS (=Visual Analog Scale) | every 3 or 4 weeks during 12 to 16 weeks
To evaluate the use of analgesic (analgesic score) and the number of patients needing an analgesic radiotherapy between V1 and V5 | every 3 or 4 weeks during 12 to 16 weeks
To evaluate the duration of responses | at 12 weeks or at 16 weeks (end of treatment)
To evaluate the number of skeletal related events by patient | every 3 or 4 weeks during 12 to 16 weeks
To evaluate the effect on functional disability, professional activity (BPI), the PS and overall condition (VAS) between V1 and V5 | every 3 or 4 weeks during 12 to 16 weeks
To evaluate the variations of PSA (=Prostate specific Antigen) between V1 and End of study or premature withdrawal | at 12 weeks or at 16 weeks (end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Monpellier, France